CLINICAL TRIAL: NCT05684341
Title: Prospective Comparison of Connected Solution (Health2Sync) and Usual Care in Adult Participants With Type 2 Diabetes Mellitus Using Basal Insulin in Taiwan
Brief Title: A Randomized Controlled Trial to Compare the Glycemic Control, With or Without the Connected Solution, of Adult Type 2 Diabetic Participants on Basal Insulin in Taiwan
Acronym: TW CES RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIR17344; U1111-1266-5860 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Intervention arm (Experimental): Connected Solution with H2S app which connects with blood glucose meter (BGM) to support glycemic control in T2DM participants
  Interventions: Combination Product: Connected Solution with H2S app which connects with blood glucose meter (BGM)
- No Device Control arm (No Intervention): Physician-recommended routine management (usual care) to support glycemic control in T2DM participants

INTERVENTIONS:
Combination Product: Connected Solution with H2S app which connects with blood glucose meter (BGM) — Combination of the Insultrate titration module software, the H2S app for participants, and the H2S platform for healthcare professionals
  Arms: Device Intervention arm

SUMMARY:
The Connected Solution investigated in this study is the combination of the titration module "Insultrate" and a cell phone application (app) named Health2Sync (H2S) that synchronizes participants' self-monitoring blood glucose data and electronic health records to a platform overseen by their treating physicians. This study investigates if this Connected Solution helps to improve glycemic control more effectively than physician-recommended routine management (i.e., usual care) in participants with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
Study duration per participant will be up to 9 months, including a screening period of up to 3 months and a study intervention period of 24 weeks (± 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 20 years of age at the time of signing the informed consent
* Participants were diagnosed with T2DM prior to the screening visit
* Participants who are insulin naïve, or already treated with basal insulin but uncontrolled with the same insulin regimen for at least 3 months (90 days) prior to Day 1
* Participants with HbA1c between 7.5% and 11% (inclusive) at the screening visit and Day 1
* Participants with fasting self-measured blood glucose (fSMBG) or fasting plasma glucose (FPG) >130 mg/dL at the screening visit and Day 1
* Capable of giving signed informed consent
* Willing and able to use the H2S app and glucometer

Exclusion Criteria:

* Participants with diabetes other than T2DM
* H2S app/ BGM is not appropriate for the participant or use of device is otherwise contraindicated (in the opinion of the investigators)
* Participants with hypoglycemia unawareness or with severe hypoglycemia within the past 90 days prior to the screening visit and until Day 1
* Hospitalization (for any reason) in the past 30 days prior to the screening visit and until Day 1
* Participants with severe conditions/concomitant diseases precluding their safety or ability to participate in this study, as judged by the investigators - Participants are not on stable dose of glucose lowering therapy including OADs, glucagon-like peptide-1 (GLP-1) receptor agonists, or basal insulin therapy within the past 12 weeks prior to the screening visit and until Day 1 per investigator's discretion
* Participants using mealtime insulin for more than 10 days in the last 90 days before the screening visit and until Day 1
* Participants who used H2S app within 1 month prior to the screening visit and until Day 1 randomization
* Participants who have taken other investigational drugs within 90 days or 5 half-lives prior to screening or randomization, whichever is longer

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at Week 24 | Baseline to Week 24

SECONDARY OUTCOMES:
Change from baseline in fasting (morning premeal) SMBG (fSMBG) at Week 24 | Baseline to Week 24
Time to first reach the fSMBG target range | Baseline to Week 24
  The time to first fSMBG reaching target range of 80 to 130 mg/dL (inclusive) will be defined as the time interval from Day 1 to the first date of reaching the target fSMBG
Insulin compliance at Week 12 and 24 | Baseline to Week 12 and 24
  Compliance (%) = (the total days of participants with insulin injecting as prescribed regimen / the total days of prescribed regimen)*100%
Insulin discontinuation rate at Week 12 and 24 | Week 12 and 24
  Percentage of participants who are discontinued from the insulin injection at Week 12 and 24
Change from baseline in total daily insulin dose at Week 12 and 24 | Baseline to Week 12 and 24
Change from baseline in body weight at Week 12 and 24 | Baseline to Week 12 and 24
Change from baseline in the score of Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) at Week 12 and 24 | Baseline to Week 12 and 24
Scores of the Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) at Week 24 | Week 24
Change from baseline in the score of the European Quality of Life 5-Dimensions 3-Level Version (EQ-5D-3L) at Week 12 and 24 | Baseline to Week 12 and 24
Number of participants experiencing hypoglycemia | Baseline to Week 24
  The number of participants experiencing hypoglycemia during the 24-week study period will be listed by threshold (glucose blood level ≤70 and <54 mg/dL) and by time window (nocturnal [00:00 to 05:59] and any time), where available
Number of hypoglycemic events per patient-year during the 24-week study period | Baseline to Week 24
  The hypoglycemic events will be listed by threshold (glucose blood level ≤70 and <54 mg/dL) and by time window (nocturnal [00:00 to 05:59] and any time), where available
Emergency room (ER) visits or hospitalizations due to hypoglycemia event | Baseline to Week 24
  Percentage of participants with at least one ER visit or hospitalization record due to hypoglycemia event per the judgment of investigators
Insulin compliance at Week 12 and 24 | Week 12 and 24
  Compliance (%) = (the total days of participants with insulin injecting as prescribed regimen / the total days of prescribed regimen)*100%
Number of participants experiencing hypoglycemia during the 24-week study period | Baseline to Week 24
  The number of participants will be listed by threshold (glucose blood level ≤70 and <54 mg/dL) and by time window (nocturnal [00:00 to 05:59] and any time), where available
Percentage of participants with at least one emergency room (ER) visit or hospitalization record due to hypoglycemia event during the 24-week study period | Baseline to Week 24
Number of participants with adverse events during the 24-week study period | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- Taiwan (14):
  - Changhua Christian Hospital - Investigational Site Number: 1580016, Changhua
  - Kaohsiung Veterans General Hospital - Investigational site number 1580010, Kaohsiung City
  - Far-Eastern Memorial Hospital - Investigational Site Number: 1580004, New Taipei City
  - Shuang Ho Hospital - Investigational Site Number: 1580012, New Taipei City
  - Chang-Gung Memorial Hospital Linkou Branch - Investigational Site Number: 1580005, New Taipei City
  - Chung-Shan University Hospital - Investigational Site Number: 1580003, Taichung
  - Tungs' Taichung Metroharbor Hospital - Investigational Site Number:1580011, Taichung
  - National Cheng Kung University Hospital - Investigational Site Number: 1580008, Tainan
  - Chi-Mai Medical Center - Investigational Site Number: 1580002, Tainan
  - National Taiwan University Hospital - Investigational site number 1580001, Taipei
  - Cathay General Hospital - Investigational Site Number: 1580006, Taipei
  - Taipei Veterans General Hospital - Investigational Site Number: 1580015, Taipei
  - Tri-Service General Hospital - Investigational Site Number: 1580014, Taipei
  - Wan Fang Hospital - Investigational Site Number: 1580013, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org